CLINICAL TRIAL: NCT03135171
Title: A Phase 1 Multi-Center Trial of Trastuzumab and Pertuzumab in Combination With Tocilizumab in Subjects With Metastatic HER2 Positive Breast Cancer Resistant to Trastuzumab
Brief Title: Trastuzumab and Pertuzumab in Combination With Tocilizumab in Subjects With Metastatic HER2 Positive Breast Cancer Resistant to Trastuzumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.002; HUM00125505 (Other: University of Michigan Comprehensive Cancer Center)
Record Dates: First submitted 2017-04-25; First posted 2017-05-01 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trastuzumab, Pertuzumab and Tocilizumab (Experimental)
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Trastuzumab — All dose levels will receive 8 mg/kg loading dose for cycle 1, followed by 6 mg/kg in subsequent cycles, every 3 weeks.
Drug: Pertuzumab — Dose Levels two and three will receive 840 mg loading dose for cycle 1, followed by 420 mg in subsequent cycles, every 3 weeks.
Drug: Tocilizumab — Tocilizumab 4-8 mg/kg, administered intravenously every three weeks

SUMMARY:
The goal in this Phase 1 dose-escalation trial of the anti-IL-6R monoclonal antibody tocilizumab in combination with trastuzumab and pertuzumab in subjects with metastatic HER2 positive breast cancer is to determine the safety, tolerability and recommended Phase 2 dose of tocilizumab given with trastuzumab and pertuzumab every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women or men with histologically confirmed breast cancer that overexpresses HER2 (defined by ASCO-CAP 2013 guidelines performed using FDA-approved tests by laboratories with demonstrated proficiency) that is metastatic or unresectable
* Subjects must have received trastuzumab in the metastatic setting and experienced disease progression on this drug.
* Any number of prior therapies is permitted. Prior therapy with other HER2 targeted agents (TDM-1, pertuzumab, lapatinib) is allowed.
* The last dose of chemotherapy must have occurred ≥3 weeks prior to study registration.
* The last radiation therapy must have occurred ≥3 weeks prior to study registration.
* Age≥ 18 years
* Eastern Cooperative Oncology Group Performance Status of 0 or 1 (An attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death.)
* Measurable and/or non-measureable disease by RECIST criteria must be present.
* Adequate organ and bone marrow function
* Subjects with treated brain metastases are eligible provided the metastases are clinically stable and greater than 8 weeks has elapsed from time of treatment and date of initiation of study drug.
* Males and females of reproductive potential must use two forms of effective contraception during the duration of the trial and for minimum of 7 months after last dose of tocilizumab, trastuzumab, or pertuzumab.

Exclusion Criteria:

* Intolerance to previous trastuzumab or pertuzumab therapy
* Previous treatment with tocilizumab or other cytokine-targeted biologic disease modifying antirheumatic drugs (including adalimumab, certolizumab, etanercept, golimumab, infliximab, anakinra) within 3 months of enrollment
* Participation in other investigational studies concurrently if these therapies include a therapeutic intervention
* Treatment with any investigational agent within 30 days (or 5 serum half-lives of the investigational drug, whichever is longer) of enrollment
* Concurrent second malignancy or history of HER2 negative breast cancer within five years
* Comorbidity or intercurrent illness
* Major surgery within 8 weeks or planned major surgery during study and up to 6 months after discontinuation of study drug
* Left ventricular systolic dysfunction, defined as ejection fraction below institutional normal by echocardiography or MUGA (multigated acquisition scan); current or past clinical diagnosis of congestive heart failure; history of ejection fraction decreased to below institutional normal or desease of greater than 15% attributable to past trastuzumab or pertuzumab therapy
* Evidence of current serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease.
* History of diverticulitis, diverticulosis requiring antibiotic treatment or chronic ulcerative lower GI (gastrointestinal) disease such as Crohn's disease, ulcerative colitis or other symptomatic lower GI conditions that might predispose to perforations
* Infections as detailed in the protocol
* Immunization with a live/attenuated vaccine within 30 days of enrollment
* Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation
* Pre-existing CNS (Central Nervous System) demyelination or seizure disorders
* Any medical or psychological condition that in the opinion of the principal investigator would interfere with safe completion of the trial
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Recommended Phase II Dose of Tocilizumab | 10 weeks
  The primary objective is to determine the highest dose level of tocilizumab (up to 8 mg/kg every 3 weeks) that, when given in combination with trastuzumab and pertuzumab every three weeks in subjects with HER2 positive metastatic breast cancer, will result in less than 25% incidence of DLT. DLTs (Dose Limiting Toxicity) will be assessed within the first two cycles (up to 10 weeks) and defined as any toxicity of grade 3 or 4, unless specifically described in the protocol.

SECONDARY OUTCOMES:
The Frequency of Adverse Events at Each Dose Level | 30 days after last treatment dose
  The number of grade 3 and 4 adverse events at each dose level will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Burness, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Yale University, New Haven, New York

IPD SHARING:
Plan to Share IPD: Undecided